CLINICAL TRIAL: NCT04100655
Title: A Randomized Controlled Trial of the Effect of the Granulocyte-macrophage Colony Stimulating Factor Gel on the Endometrial Thickness in Infertile Women With Thin Endometrium
Brief Title: The Effect of the GM-CSF Gel on the Endometrial Thickness in Infertile Women With Thin Endometrium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiaona Lin, Vice Director of gynaecology and obstetrics, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRRSH20190806-19
Record Dates: First submitted 2019-09-03; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Thin Endometrium
Keywords: GM-CSF; frozen embryo transfer
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; femoston

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GM-CSF (Experimental): Hysteroscopy will be arranged to confirm the uterine cavity is normal and there is no significant intrauterine adhesion.
  3ml GM-CSF gel will be irrigated into the uterine cavity immediately when hysteroscopy is complete. Then same dose gel will be given every other day twice.
  Interventions: Drug: GM-CSF; Drug: 17-ß estradiol
- Control (Experimental): Hysteroscopy will be arranged to confirm the uterine cavity is normal and there is no significant intrauterine adhesion.
  After hysteroscopy examination, nothing was applied to the uterine cavity.
  Interventions: Drug: 17-ß estradiol

INTERVENTIONS:
Drug: GM-CSF — 3ml GM-CSF gel will be irrigated into the uterine cavity immediately when hysteroscopy is complete. Then same dose gel will be given every other day twice
  Other Names: granulocyte-macrophage colony stimulating factor
  Arms: GM-CSF
Drug: 17-ß estradiol — A hormone replace treatment by 17-ß estradiol (6mg per day) follows next cycle to prepare for embryo transfer
  Other Names: Femoston

SUMMARY:
The purpose of this study is to investigate the efficacy of the granulocyte-macrophage colony stimulating factor(GM-CSF) gel on the endometrial thickness in infertile women with thin endometrium.

DETAILED DESCRIPTION:
The thin endometrium is detrimental to embryo implantation, probability of clinical pregnancy for an endometrial thickness ≤ 7 mm was significantly lower compared with cases with endometrial thickness > 7 mm. It has been reported the granulocyte colony stimulating factor (G-CSF) increased the endometrial thickness and pregnancy rate of infertile women with thin endometrium during IVF cycle. However, most of the researches were retrospective and small sample size, and the results were conflicted among them. GM-CSF is another member of CSF superfamily, recalling more macrophage than G-CSF, which could be more effective in local homeostasis maintain and wound repair. GM-CSF has been widely used in skin repair after burn. It was also found the GM-CSF and its receptor in endometrium. In the past year, the investigators tried GM-CSF irrigation in 21 women with thin endometrium and most of them received GM-CSF after hysteroscopic examination or slight adhesion relaxing, and the preliminary data suggested that the GM-CSF may promote the endometrial growth. Does the GM-CSF gel can improve the endometrial thickness? Therefore, this study was conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Woman undergoes IVF treatment, 18-40 years old
2. The endometrial thickness <7mm on the day of human chorionic gonadotropin during IVF or after taking oral estradiol valerate 6mg/d for 14 days.
3. Embryo transfer is cancelled because of thin endometrium
4. No intrauterine adhesion according to the 3-D ultrasonography

Exclusion Criteria:

1. Systemic diseases unable to conceive
2. Chromasome abnormal
3. History of G-CSF or GM-CSF allergy or untoward effect
4. Thin endometrium related to clomid
5. Severe or moderate uterine adhesion
6. The influence factor of embryo implantation: hydrosalpinx, endometriosis, adenomyosis,myoma of uterus
7. Uterine malformation, adenomyosis, uterine leiomyoma sized more than 2cm.
8. Patients who is allergic to granulocyte-macrophage colony stimulating factor
9. Patients with inflammation of reproductive organs, pelvic cavity inflammation, malignant tumor of reproductive organs and other systemic diseases that could cause metrorrhagia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
the endometrial thickness | 1 months after hysteroscopy examination
  the endometrial thickness following the hormonal replacement treatment evaluated based on the ultrasound

SECONDARY OUTCOMES:
embryo transfer cancelation rate | 2 months after hysteroscopy examination
  according to the patients' wishes
uterine artery blood supply markers | 1 months after hysteroscopy examination
  uterine artery blood supply markers, such as PI, reflux index(RI) and S/D, evaluated based on the 3-D ultrasonography
pregnancy rate | 3 months after hysteroscopy examination
  pregnancy rate after frozen embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Xiaona Lin, Doctor, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No